CLINICAL TRIAL: NCT06807515
Title: Pilot Observational Study and Safety Analysis of FL Nourish Capsules in Cancer Patients in Remission
Status: Enrolling by invitation | Type: Observational
Sponsor: Thong Chai Institute of Medical Research (Other)
Responsible Party: Sponsor
Other Study IDs: TCIMR-FLNC1
Record Dates: First submitted 2025-01-22; First posted 2025-02-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Cancer Survivor
Keywords: cancer; herbal medicine; traditional chinese medicine; chinese herbal medicine; tcm; complementary; alternative; fatigue; Cancer-related fatigue
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FLNC Group

SUMMARY:
This is a single-centre, observational prospective study of cancer patients in remission administering FL Nourish capsules (FLNC), a proprietary Chinese Medicine herbal supplement, for the treatment of symptoms associated with qi deficiency and blood stasis syndrome.

DETAILED DESCRIPTION:
Consultation data will be analysed from up to 24 cancer patients in remission receiving routine treatment at Singapore Thong Chai Medical Institution. Each participant will visit the institution in accordance with the protocol which includes up to 9 months of FL Nourish capsule (FLNC) use and up to 8 consultation visits. Participants will be evaluated based on consultation data, questionnaire data, routine blood test data and self-reporting of adverse events or severe adverse events. As this is a non-interventional observational study, all participants would have received FLNC prescriptions according to routine diagnostic and prescribing standards, and there were no additional visits required aside from routine follow up consultations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-80;
* Cancer diagnosis ≤ 5 years;
* Received treatment with no current evidence of recurrence, with predicted life expectancy of 12 months and above;
* On regular follow-up with lab tests scheduled every 1-9 months;
* Recent (<=3 months) blood test report(s) available on first study visit
* Diagnosed with the TCM syndrome of Qi deficiency and Blood stasis by the primary physician: experience 2 major symptoms coupled with typical tongue and pulse conditions; 2 major symptoms and 1 possible symptom coupled with tongue and pulse conditions; and 1 major symptom and at least 2 possible symptoms coupled with tongue and pulse conditions;

Exclusion Criteria:

* On active cancer treatment such as IV chemotherapy or radiotherapy or oral targeted therapy (excluding HRT and oral chemotherapy);
* Scheduled for IV chemotherapy, radiotherapy or surgery within the next 1 year from recruitment date;
* Diagnosed with active disease of the liver, kidney, brain, blood, blood vessels; with mental health conditions or are mentally incapacitated;
* Pregnant women.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical stable, post-treatment cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-02-09 (Estimated); Study Completion 2027-08-09 (Estimated)

PRIMARY OUTCOMES:
Pre-post values of EORTC QLQ-C30 questionnaire test scores | From enrollment to the end of treatment at 10 months
  0 is equivalent to a low QoL/functioning/symptom score and 100 indicates the best posssible QoL/functioning/symptom score.

SECONDARY OUTCOMES:
Incidence of unanticipated adverse events or severe adverse events: estimated to be <= 10% | From enrollment to the end of treatment at 10 months
Pre-post values of Alanine aminotransferase (ALT) | From enrollment to the end of treatment at 10 months
Pre-post values of Aspartate aminotransferase (AST) | From enrollment to the end of treatment at 10 months
Pre-post values of albumin-to-creatinine ratio (ACR) | From enrollment to the end of treatment at 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Huang Fang Zheng, PhD, BS, Study Director — Singapore Thong Chai Medical Institution; Renyuan Shen, MS, BA, Principal Investigator — Singapore Thong Chai Medical Institution
Locations (1):
- Singapore Thong Chai Medical Institution, Singapore, SG, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan A, Chan D, Ng DQ, Zheng HF, Tan QM, Tan CJ, Toh JHM, Yap NY, Toh YL, Ke Y, Wang ECA, Lim QPN, Ho HK, Chew L, Tan TJ. HEalth-Related Quality of Life-Intervention in Survivors of Breast and Other Cancers Experiencing Cancer-Related Fatigue and Associated Cognitive Symptoms Using TraditionAL Chinese Medicine: The 'HERBAL' Trial. Integr Cancer Ther. 2025 Jan-Dec;24:15347354251314514. doi: 10.1177/15347354251314514. PMID 39840742